CLINICAL TRIAL: NCT07008183
Title: Perinatal Thymic Dysregulation: Characterization of Perinatal Mood Episodes
Acronym: DYP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A02708-39; ID-RCB (Other: ANSM)
Record Dates: First submitted 2025-05-06; First posted 2025-06-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Perinatal Mental Health
Keywords: perinatal mental health; perinatal depression; perinatal bipolar troubles

STUDY DESIGN:
Intervention Model Description: Participants are assigned prospectively to complete self-questionnaires according to the protocol to characterize perinatal mood episodes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual care (Experimental): The study aims to systematize the evaluation of the various criteria used to characterize mood episodes, and to explore contextual elements.
  Interventions: Other: self-questionnaires

INTERVENTIONS:
Other: self-questionnaires — Patients who volunteer to take part in the research will complete self-questionnaires before their appointment with the psychiatrist.

SUMMARY:
The perinatal period is recognized as a time of heightened psychological vulnerability. This research aims to improve the diagnosis and therapeutic management of mood episodes occurring during this time. It is integrated into routine clinical care and seeks to standardize the evaluation of criteria used to characterize mood episodes, while also exploring relevant contextual factors.

Traditionally, clinical attention has focused on postnatal depression; however, increasing evidence highlights the presence of hypomanic symptoms-such as distractibility, reduced need for sleep, tachypsychia, and irritability-during the postpartum period. These symptoms may coexist with depressive features, resulting in complex clinical presentations that are often difficult to recognize and manage. Consequently, many cases go undiagnosed and untreated.

Current research has largely concentrated on depressive episodes (perinatal depression), with less emphasis on manic, hypomanic, or mixed episodes indicative of bipolar disorder. A systematic evaluation of hypomanic symptoms occurring alongside depressive symptoms in the postpartum period could refine clinical diagnosis and support more targeted and effective therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Pregnant or having given birth less than a year ago
* First psychiatric consultation for the pregnancy concerned.
* Good command of the French language.
* Participant affiliated to the social security system
* Participant who has given her consent to take part in the study.

Exclusion Criteria:

* Women who gave birth more than a year ago.
* Participant under psychiatric care
* Participant under court protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detailed description of the Edinburg Postnatal (EPDS) scale | 1 day
  A sensitivity analysis will be carried out on the group of patients with an EPDS score greater than 12, and a comparison between these patients and patients with an EPDS score equal to or less than 12 will also be carried out
Detailed description of Multidimensional Assessment of Thymic (MAThyS) scale | 1 day

SECONDARY OUTCOMES:
Association of the risk factors Perceived Stress Scale (PSS) will be assessed by self-report | 1 day
  the level of perceived stress by self report score>=14 characterize a high level of perceived stress
Association of the risk factors Medical Outcomes Study -Social Support Survey (MOS-SSS) will be assessed by self-report | 1
  the level of perceived social support by self-report scale scores can range from 19 to 95, with a median score of 57
Association of the risk factors Perceived Professional Social Support (QSSP-P) will be assessed by self-report | 1
  the level of perceived social support in the professional by self-report. scale scores pcan range from 12 to 120, with a median score of 66

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure SUTTER-DALLAY, Prof Md PhD, Principal Investigator — Centre Hospitalier Charles Perrens
Locations (1):
- Centre Hospitalier CHARLES PERRENS, Bordeaux, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beck CT. Predictors of postpartum depression: an update. Nurs Res. 2001 Sep-Oct;50(5):275-85. doi: 10.1097/00006199-200109000-00004. PMID 11570712
- [Result] Ballinger CB. Emotional disturbance during pregnancy and following delivery. J Psychosom Res. 1982;26(6):629-34. doi: 10.1016/0022-3999(82)90079-4. PMID 7161736
- [Result] Areias ME, Kumar R, Barros H, Figueiredo E. Correlates of postnatal depression in mothers and fathers. Br J Psychiatry. 1996 Jul;169(1):36-41. doi: 10.1192/bjp.169.1.36. PMID 8818366
- [Result] Appleby L. Suicide during pregnancy and in the first postnatal year. BMJ. 1991 Jan 19;302(6769):137-40. doi: 10.1136/bmj.302.6769.137. PMID 1995132
- [Result] Anderson D, Bilodeau B, Deshaies G, Gilbert M, Jobin J. [French-Canadian validation of the MOS Social Support Survey]. Can J Cardiol. 2005 Aug;21(10):867-73. French. PMID 16107910